CLINICAL TRIAL: NCT05844033
Title: Biomarker for Infection Risk in Chronic Lymphocytic Leukemia and Multiple Myeloma
Brief Title: Biomarker for Infection Risk in CLL and MM
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Jacob Soumerai, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 23-105
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: Multiple Myeloma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Antibody profiling and functional assays (advanced testing which detects antibodies directed against specific pathogens and measures their functional capacity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia and Multiple Myeloma Participants: 150 participants will be screened for an antigen-specific antibody profiling biomarker that is associated with an increased risk of any infections.
  Study procedures include in-person or virtual appointments every 3 months for 2 years, some of which will also include bloodwork:
  * In-person or virtual appointments with study staff for months 4, 10, 16, and 22 Day 1.
  * In-person or virtual appointments with study staff for months 7, 13, 19, and 25 Day 1 with blood tests.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Blood tests

SUMMARY:
The aim of this research study is to use advanced immunology laboratory analysis to identify a more precise blood test that will predict infection risk in patients with Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma (CLL/SLL) or Multiple Myeloma (MM).

DETAILED DESCRIPTION:
The goal of this research study is to identify an antigen-specific antibody profiling biomarker associated with increased risk of any infections in patients with Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma (CLL/SLL) or Multiple Myeloma (MM).

Research procedures including screening for eligibility, clinic visits, and blood tests.

This involves performing blood tests which detect antibodies directed against specific pathogens and measure their functional capacity, and collecting information about outcomes in patients.

Participation in this research study is expected to last 2 years.

It is expected that about 150 people CLL or MM will take part in this research study, and this will predominantly include people with CLL/SLL.

Takeda is supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Diagnosis of Rai stage I-IV chronic lymphocytic leukemia or small lymphocytic lymphoma or multiple myeloma.
* Subjects must be able to consent to clinical trial, or documented health care proxy agent able to consent on behalf of participant.

Exclusion Criteria:

* Subjects must not have received IVIG administration within 6 calendar months of registration or have planned immunoglobulin replacement therapy by treating investigator at time of registration.
* Subjects with chronic lymphocytic leukemia or small lymphocytic lymphoma must not be Rai stage 0.
* Subjects with multiple myeloma must not have smoldering myeloma or solitary plasmacytoma with or without minimal marrow involvement.
* Subjects must not have undergone prior autologous, allogeneic stem cell, or solid organ transplant.
* Subjects must not have any active systemic infection requiring ongoing antimicrobial treatment (prophylactic antimicrobial allowed) at time of registration.
* Subjects must have no known history of HIV, primary immune deficiency disorder, nor be taking a concurrent immune suppressing medication at time of registration. Treatment for CLL/SLL or MM, CLL/SLL related autoimmune phenomenon, or physiologic dosing of corticosteroids (5mg/day prednisone/equivalent or lower) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnoses of Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Multiple Myeloma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of All-Grade Infections For All Participants | up to 2 years
  Defined as the number of All-Grade infections per person-years per CTCAE version 5.0 for all participants.

SECONDARY OUTCOMES:
Number of Grade ≥3 Infections For All Participants | up to 2 years
  Defined as the number of Grade ≥3 infections per person-years per CTCAE version 5.0 for all participants.
Number of All-Grade Infections for Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Leukemia (SLL) Participants | Up to 2 years
  Defined as the number of All-Grade infections per person-years per CTCAE version 5.0 for CLL/SLL participants.
Number of Grade ≥3 Infections for Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL) Participants | up to 2 years
  Defined as the number of Grade ≥3 infections per person-years per CTCAE version 5.0 for CLL and SLL participants.
Number of All-Grade Infections for Multiple Myeloma (MM) Participants | up to 2 years
  Defined as the number of All-Grade infections per person-years per CTCAE version 5.0 for MM participants.
Number of Grade ≥3 Infections for Multiple Myeloma (MM) Participants | up to 2 years
  Defined as the number of Grade ≥3 infections per person-years per CTCAE version 5.0 for MM participants.
Proportion of patients who develop symptomatic hypogammaglobulinemia in CLL/SLL or MM. | Up to 2 years
  Defined as any incident in which immunoglobulin replacement therapy is administered to an participant who develops symptomatic hypogammaglobulinemia with Immunoglobulin G <600mg/dL and either 1) ≥2 associated infections within a 6-month period, or 2) any grade ≥3 associated infection.
Proportion of patients who develop asymptomatic hypogammaglobulinemia in CLL/SLL or MM. | Up to 2 years
  Defined as the proportion of all participants who develop symptomatic hypogammaglobulinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Soumerai, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation.